CLINICAL TRIAL: NCT02769650
Title: Clinical Significance of Stress-MRI Evaluation of Right Coronary Artery Chronic Total Occlusion Recanalization Efficacy in Patients With Coronary Artery Disease.
Brief Title: Stress-MRI Assessment After Right Coronary Artery CTO Recanalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Stress-MRI 1.0
Record Dates: First submitted 2016-05-08; First posted 2016-05-11 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Ischemic Heart Disease; Coronary Atherosclerosis; Coronary Artery Disease; Coronary Artery Stenosis
Keywords: Coronary stenosis; Drug-eluting stent; Coronary angioplasty with stenting; Ischemic Heart Disease; Chronic total occlusion; Right coronary artery; Stress-MRI
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stress-MRI + Chronic total occlusion PCI (Experimental): Pre- and postoperative stress-MRI with evaluation of myocardium perfusion defects + Coronary angioplasty with stenting of RCA CTO
  Interventions: Procedure: CTO coronary angioplasty; Procedure: Stress-MRI
- Stress-MRI + Optimal medicamentous treatment (Active Comparator): Pre- and postoperative stress-MRI with evaluation of myocardium perfusion defects + Optimal medicamentous treatment
  Interventions: Drug: Optimal medicamentous treatment; Procedure: Stress-MRI

INTERVENTIONS:
Procedure: CTO coronary angioplasty — A standard endovascular procedure is carried out under local anesthesia and under fluoroscopic control. Recanalisation of coronary artery CTO is performed by the hydrophilic coronary wire, using the most appropriate technique. Then balloon angioplasty of target lesion is provided. After the angiographic control coronary stent is implanted. After coronary wire removing control angiographic study is provided. Medical therapy includes aspirin(acid acetylsalicylic) 125 - 300 mg/d and plavix(clopidogrel) in dose 300-600 mg prescription before the procedure and heparin (heparin sodium) injection during the procedure(5000 U iv). After the procedure aspirin(acid acetylsalicylic) in dose 100 mg/d within long period should be prescribed in all the patients, and plavix(clopidogrel) in dose 75/d should be prescribed within 12 months.
  Arms: Stress-MRI + Chronic total occlusion PCI
Drug: Optimal medicamentous treatment
  Arms: Stress-MRI + Optimal medicamentous treatment
Procedure: Stress-MRI — A standard stress-MRI test with adenosine

SUMMARY:
The hypothesis of this study is that Stress-MRI is a clinically significant method of myocardial perfusion assessment after coronary angioplasty with stenting of right coronary artery (RCA) chronic total occlusion (CTO) is performed.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina, CCS FC II-IV
* "Right-dominance" coronary circulation according to coronary angiography
* Absence of other significant atherosclerotic coronary lesions (more than 65%)
* High risk of myocardium ischemia according to stress-MRI data (perfusion defect in 2 or more segments in the area of interest)
* Signed, documented informed consent prior to admission to the study

Exclusion Criteria:

* Acute coronary syndrome
* Contraindications for adenosine stress test
* Low and moderate risk of myocardium ischemia according to stress-MRI data (perfusion defect in less than 2 segments in the area of interest)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Stress-MRI evaluation | Within 2 and 12 month after hospitalization
  High risk of myocardium ischemia according to stress-MRI data (perfusion defect in 2 or more segments in the area of interest)

SECONDARY OUTCOMES:
Clinical assessment | Within 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 moths after hospitalization
  Dynamical assessment of stable angina FC (CCS) and dyspnea FC (NYHA)
Stress-MRI evaluation (2) | Within 2 and 12 month after hospitalization
  Dynamics of perfusion in myocardium scar tissue according to stress-MRI data
Major adverse cardiac and cerebrovascular events (MACCE) | During 1 year after first stress-MRI assessment
  Major adverse cardiac and cerebrovascular events (MACCE) including: All-cause mortality, Myocardial infarction, Stroke, Stent thrombosis, Clinically indicated Target lesion revascularization, Any target lesion revascularization, Any target vessel revascularization.

CONTACTS AND LOCATIONS:
Locations (1):
- State Research Institute of CIrculation Pathology, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No